CLINICAL TRIAL: NCT00000201
Title: Pharmacological Modulation of Cocaine Effects
Brief Title: Pharmacological Modulation of Cocaine Effects - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Johns Hopkins University (Other)
Purpose: Treatment
Other Study IDs: NIDA-05196-1; R01-05196-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Selegiline

INTERVENTIONS:
Drug: Selegiline

SUMMARY:
The purpose of this study is to conduct human laboratory studies of possible cocaine interactions with various potential treatment medications.

ELIGIBILITY:
Please contact site for information.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0
Dates: Study Completion 2001-12

CONTACTS AND LOCATIONS:
Overall Officials: George Bigelow, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University (BPRU) Bayview Campus, Baltimore, Maryland, United States